CLINICAL TRIAL: NCT04158167
Title: Neurobiological Effects of Oxytocin on Metacognitive Deficits in Schizophrenia: A Pharmacological - Imaging Genetics Study
Brief Title: Neurobiological Effects of Oxytocin in Schizophrenia - Imaging Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Dr Naren P Rao, Additional Professor, National Institute of Mental Health and Neuro Sciences, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00807
Record Dates: First submitted 2019-11-01; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: After completion of clinical and cognitive assessments, all subjects will undergo a baseline fMRI scan. Later subjects will receive24IU oxytocin and saline placebo in counterbalanced order on two separate days and undergo repeat fMRI scans.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- oxytocin (Other): All subjects will receive both oxytocin and placebo in a counterbalanced design
  Interventions: Drug: oxytocin

INTERVENTIONS:
Drug: oxytocin — 24 International units of oxytocin or palcebo will be given intranasally. The order of administration will be counterbalanced

SUMMARY:
To investigate whether 24IU oxytocin can result in changes in functional brain connectivity in patients with schizophrenia and healthy individuals using functional magnetic resonance imaging (fMRI). The study will also examine the effect of oxytocin receptor gene polymorphism on the functional connectivity

ELIGIBILITY:
Inclusion and Exclusion Criteria:

Schizophrenia subjects:

Inclusion criteria 1) Males between 18 and 50 years 2) Diagnosis of DSM-IV schizophrenia, schizoaffective or schizophreniform disorder 3) capacity to provide informed consent, as evaluated by the MacArthur Competence Assessment Tool for Clinical Research Exclusion criteria

1. General impairment in intellectual functioning
2. History of alcohol or substance dependence in the last 12 months (with the exception of nicotine)
3. Contraindication to oxytocin like hypersensitivity, vascular disease, chronic nephritis, epilepsy, asthma
4. Past history of head injury resulting in loss of consciousness or neurosurgery
5. Concomitant severe medical conditions
6. Metal implants or paramagnetic objects within the body or claustrophobia which may interfere with the MRI.

Healthy volunteers:

Inclusion criteria

1. Males between 18 and 50 years
2. Capacity to provide informed consent Exclusion criteria

1) Life-time diagnosis of psychiatric illnesses including substance abuse 2) General impairment in intellectual functioning 3) Past history of head injury resulting in loss of consciousness or neurosurgery 4) Concomitant severe medical or neurological conditions 5) Metal implants or paramagnetic objects or claustrophobia 6) Family history of schizophrenia, schizoaffective or schizophreniform disorder in family member (sibling, parent or offspring) 7) Contraindication to oxytocin like hypersensitivity, vascular disease, chronic nephritis, epilepsy, asthma.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
fMRI changes with oxytocin | Upto 90 minutes after administration
  changes in functional brain connectivity

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health and Neurosciences, Bangalore, Karnataka, India